CLINICAL TRIAL: NCT07183995
Title: Hematological Disorders in Patients With Gastrointestinal Angiodysplasia
Brief Title: Hematological Disorders in Patients With GI Angiodysplasia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mennat-allah Alaa Abdelgaber Omar, Principal investigatir, Assiut University
Other Study IDs: GI angiodysplasia patients
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: GI Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study will be to assess the association between GIT angiodysplasia with any hematological disorders as von Willebrand factor and Prognostic value of von Willebrand factor on patient's outcomes as risk of rebleeding and hospital mortality

ELIGIBILITY:
Inclusion Criteria:

Adults (above 18 years) and elderly Both genders Admitted to GIT Unit with manifestations of GIT bleeding diagnosed by upper endoscopy and Colonoscopy as angiodyplasia.

-

Exclusion Criteria:

other causes of GIT bleeding

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients eligible to participate will undergo the following:
  1. upper endoscopy
  2. Colonoscopy
  3. Complete blood count, CRP
  4. D-Dimer, liver function tests, blood Urea and serum Creatinine
  5. ECG
  6. Coagulation profile (aPTT , von Willebrand factor activity &antigen)
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Correlation between GIT Angiodysplasia and Hematological disorders | Baseline
  All patients eligible to participate will undergo the following:
  1. upper endoscopy
  2. Colonoscopy
  3. Complete blood count, CRP
  4. D-Dimer, liver function tests, blood Urea and serum Creatinine
  5. ECG
  6. Coagulation profile (aPTT , von Willebrand factor activity &antigen)

SECONDARY OUTCOMES:
Prevelance of different hematological disorders in angiodysplasia patients | Baseline
Prognostic value of von Willebrand factor on patient's outcomes as risk of rebleeding and hospital mortality | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mennat-allah Alaa Abdelgaber, Principal Investigator — Assiut University; Mohamed Zein Elabdin Hafez, Study Director — Assiut University; AbdelHamid Mohamed AbdelHamid, Study Director — Assiut University